CLINICAL TRIAL: NCT06981143
Title: "Investigation of Knowledge and Perceptions of Physical Activity and Exercise of Greek Specialists and Residents in Pathological Oncology"
Brief Title: Oncologists' Perceptions on Physical Activity and Exercise
Status: Completed | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Syrou Niki, RN,MPH, PhD, Laboratory Teaching Staff, University Lecturer, University of Thessaly
Other Study IDs: PAE-Oncologists' perceptions
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Perceptions on Physical Activity and Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oncologists: All Greek specialists and medical residents in pathological oncology who manage patients with cancer.
  Interventions: Behavioral: Quantitative study

INTERVENTIONS:
Behavioral: Quantitative study — A validated questionnaire will be used to investigate the knowledge and perceptions of physical activity and exercise of specialists and residents in Pathological Oncology

SUMMARY:
The aim of this observational and nationwide study is to investigate the knowledge and perceptions of the entire population of Greek specialists and medical residents in pathological oncology regarding physical activity and exercise in patients with cancer. Sub-objectives of the study are to investigate the barriers and facilitating factors in counseling and prescribing exercise in cancer patients. The data collection will be conducted through a validated questionnaire developed in a previous study, which will be sent via an online Google Form platform, ensuring the anonymity and confidentiality of the participants' responses. The questionnaire will include demographic characteristics, four basic scales with mandatory responses (subjective knowledge, attitudes, skills and behaviour in physical activity and exercise) and an optional scale of objective knowledge in physical activity and exercise.

ELIGIBILITY:
Inclusion Criteria:

* All specialists and residents in Pathological Oncology in Greece

Exclusion Criteria:

* Physicians of other specialties other than Pathological Oncology
* Greek Pathological Oncologists who practice the specialty of Pathological Oncology abroad.

Ages: 24 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Specialists and residents in Pathological Oncology in Greece.
Sampling Method: Non-Probability Sample
Enrollment: 606 (Actual)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2026-02-02 (Actual)

PRIMARY OUTCOMES:
Investigation of oncologists' perceived knowledge on physical activity and exercise via questionnaire. | Once during the study (i.e. from 05/2025 to 10/2025)
  Only physicians, specialists, and residents in pathological oncology who manage patients with cancer will be included.
  Likert-type scale questions, with responses ranging from 1 to 5 (low to high level of perceived knowledge).
  Higher scores mean a better outcome.
Investigation of oncologists' attitudes on physical activity and exercise via questionnaire | Once during the study (i.e. from 05/2025 to 10/2025)
  Only physicians, specialists, and residents in pathological oncology who manage patients with cancer will be included.
  Likert-scale questions, with responses ranging from 1 to 5 (low to high level of agreement with statements).
  Higher scores mean a better outcome.
Investigation of oncologists ' abilities to promote physical activity and exercise via questionnaire | Once during the study (i.e. from 05/2025 to 10/2025)
  Only physicians, specialists, and residents in pathological oncology who manage patients with cancer will be included.
  Likert-type scale questions, with responses ranging from 1 to 5 (low to high level of perceived ability).
  Higher scores mean a better outcome.
Investigation of oncologists ' behavior on physical activity and exercise via questionnaire | Once during the study (i.e. from 05/2025 to 10/2025)
  Only physicians, specialists, and residents in pathological oncology who manage patients with cancer will be included.
  Likert-type scale questions, with responses ranging from 1 to 5 (never to always).
  Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Investigation of oncologists' objective knowledge on physical activity and exercise via questionnaire. | Once during the study (i.e. from 05/2025 to 10/2025)
  Only physicians, specialists, and residents in pathological oncology who manage patients with cancer will be included.
  Potential responses include ''True'', ''False'', and ''Don't know''. Higher scores mean a better outcome.
Investigation of oncologists' facilitators and barriers on physical activity and exercise councelling and prescription via questionnaire | Once during the study (i.e. from 05/2025 to 10/2025)
  Only physicians, specialists, and residents in pathological oncology who manage patients with cancer will be included.
  1. Likert-type scale questions, with responses ranging from 1 to 5 (never to always). Higher score regarding facilitators means a better outcome, while a higher score regarding barriers means a worse outcome.
  2. Multiple choice questions.

CONTACTS AND LOCATIONS:
Overall Officials: Niki Syrou, PhD, Study Chair — Department of Physical Education and Sport Science, University of Thessaly; Athanasios Jamurtas, Professor, Study Chair — Department of Physical Education and Sport Science, University of Thessaly; Antonios Stavropoulos-Kalinoglou, Professor, Study Chair — Department of Physical Education and Sport Science, University of Thessaly; Evangelos Voulgaris, PhD, Principal Investigator — Department of Physical Education and Sport Science, University of Thessaly
Locations (1):
- Department of Physical Education and Sports Science, University of Thessaly, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Abstract of the European Journal of Public Health (ID: ckad160.1139), Volume 33 Supplement 2, 2023 — https://pmc.ncbi.nlm.nih.gov/articles/PMC10597221/
- See also: Postdoctoral Thesis in Repository — https://pergamos.lib.uoa.gr/uoa/dl/object/3371395